CLINICAL TRIAL: NCT01542606
Title: Performance Proof of The Norma-Sense Gen 3 - Wearing Study
Brief Title: Performance Proof of Product Developed to Detect Abnormal Vaginal pH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal decision of the sponsor
Sponsor: Common Sense (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: F-7-28.6-1
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-08

CONDITIONS: Vaginal Infection
Keywords: PH; SCREENING; EARLY WARNING; VAGINAL HEALTH; VAGINAL SECRETION; VAGINAL PH
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- color status (Experimental): The NORMA-SENSE gen 3 polymer matrix is stained by blue or green color on a pale yellow background when the pH level of the fluid in contact with it is greater than the cutoff value, and the user can consider any stain of color, which is different from the original background, as a positive result of the test.
  Interventions: Device: NORMA-SENSE

INTERVENTIONS:
Device: NORMA-SENSE — The NORMA-SENSE gen 3 polymer matrix is stained by blue or green color on a pale yellow background when the pH level of the fluid in contact with it is greater than the cutoff value, and the user can consider any stain of color, which is different from the original background, as a positive result of the test.

SUMMARY:
This study was designed to validate the color appearance on the NORMA-SENSE gen 3 when comes into contact with vaginal secretions having an elevated pH level

DETAILED DESCRIPTION:
This study was designed to validate the color appearance on the NORMA-SENSE gen 3. The NORMA-SENSE gen 3 changes color when worn by the user and comes into contact with vaginal secretions having an elevated pH level, without false positives due to urine remains or incontinence. The study will also asses the physical comfort in using NORMA-SENSE gen 3 and the result reading clarity which includes the ability to visualize and interpret the NORMA-SENSE gen 3 results.

ELIGIBILITY:
Inclusion Criteria:

1. Women, age 18 years or greater with or without symptoms of vaginal infection.
2. Subject is ready to sign the informed consent form.

Exclusion Criteria:

1. Subject is unable or unwilling to cooperate with study procedures.
2. Subject is currently participating in another clinical study.
3. Subject suffers from vaginal bleeding or is menstruating.
4. Subject that have had sexual relations within the last 12 hours.
5. Subject that applied local antiseptic or antibiotic or vaginal treatment within the last 3 days.
6. Subject that applied vaginal douching within 12 hours prior to the visit at the clinic.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
color status of the NORMA-SENSE gen 3 and the pH measurement. | 3 days
  agreement between the color status of the NORMA-SENSE gen 3 as reported by the subject after using the panty liners, and the pH measurement with Nitrazine paper.

SECONDARY OUTCOMES:
physical comfort in using NORMA-SENSE gen 3 and the result reading clarity | 3 days
  the patient report regarding physical comfort in using NORMA-SENSE gen 3 and the result reading clarity including the ability to visualize and interpret the NORMA-SENSE gen 3 results.

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Kessary, PhD, Study Director — Common Sense
Locations (1):
- Lin Medical Center Clalit health care, Haifa, Israel